CLINICAL TRIAL: NCT07323914
Title: A Clinical Study on the Efficacy of Analgesic Treatments for Chronic Pain in Patients With Dementia
Brief Title: Clinical Analgesic Management in Dementia
Acronym: CALM-D
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025005001
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; chronic pain; opioid drugs
MeSH Terms: conditions — Alzheimer Disease; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tylex group (Experimental)
  Interventions: Drug: Tylex

INTERVENTIONS:
Drug: Tylex — Tylenol (compound oxycodone/acetaminophen) is a non-narcotic analgesic that combines a lower dose of oxycodone (5 mg) with acetaminophen (325 mg). Compared to OxyContin, it provides milder opioid potency and utilizes a synergistic mechanism to achieve pain control with reduced risk of opioid-related side effects.

SUMMARY:
This study is designed to assess the efficacy and safety of oxycodone in managing moderate to severe pain in patients with Alzheimer's disease. The trial will be conducted at Xuanwu Hospital, Capital Medical University, and will enroll 10 eligible participants. Participants will receive oxycodone/acetaminophen (5 mg/325 mg) once daily for 12 weeks. The treatment will follow international guidelines, with dosages adjusted based on the patient's baseline pain levels and individual needs. Dosages will be adjusted based on baseline pain levels and patient needs, following international guidelines. Efficacy and adverse events will be assessed at baseline, week 6, week 12, and at a 12-week post-treatment follow-up. The primary outcome is change in VAS pain scores; secondary outcomes include PAINAD, SF-36, functional ability, and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 50 to 90 years at the time of enrollment.
* Meets the NIA-AA core clinical diagnostic criteria for probable Alzheimer's disease.
* Clinical Dementia Rating - Global Score (CDR-GS) between 0.5 and 2.0, inclusive, and Clinical Dementia Rating - Memory Box (CDR-MB) score ≥ 0.5.
* Diagnosed with chronic pain within 6 months prior to enrollment and considered appropriate for opioid therapy.
* Presence and severity of pain confirmed using PAINAD, MOBID-2, or comparable scales.
* Educational attainment: at least 4-6 years of formal education, or not illiterate.
* If currently receiving psychotropic or cognitive-enhancing medications, the dosage must have been stable for at least 3 months prior to study entry and remain unchanged during the study. Unless otherwise specified, all other permitted concomitant medications (non-AD related) must be stably administered for at least 4 weeks prior to baseline.
* Has a reliable caregiver/companion who can assist with study participation, defined as a person who can support the participant throughout the study and spend at least 8 hours per week with the participant.
* Willing and able to participate in this clinical trial, to maintain the assigned intervention during the study period, and has signed the informed consent form.

Exclusion Criteria:

* History of transient ischemic attack (TIA), stroke, or seizure within the past 12 months.
* Presence of any psychiatric diagnosis or symptoms that may interfere with study participation (e.g., hallucinations, major depression, or delusions).
* Known allergy to opioid analgesics.
* Severe visual or hearing impairment.
* Alcohol dependence, substance abuse, or other drug addiction or addictive tendency.
* Current participation in another study related to the treatment of Alzheimer's disease.
* Any other uncontrolled or inadequately treated medical condition (e.g., cardiac, respiratory, gastrointestinal, hepatic, or renal disease), or any condition judged by the investigator to compromise participant safety or interfere with study assessments.
* Any other reason deemed by the investigator to preclude participation in the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment in Advanced Dementia Scale (PAINAD) | baseline, 6 weeks, 12 weeks, 24 weeks.

SECONDARY OUTCOMES:
Changes from baseline of exploratory blood biomarkers | baseline; 12 weeks.
  Description: Exploratory blood biomarkers related to astrocyte-neuron interactions will be assessed using the SomaScan 11k platform. These include glial fibrillary acidic protein (GFAP), S100B, YKL-40, β-synuclein, neuregulin 1, GluN2A, and neurogranin.
Mobilization-Observation-Behavior-Intensity-Dementia Pain Scale, version 2 (MOBID-2) | baseline, 6 weeks, 12 weeks, 24 weeks.
Change from Baseline in Brain Amyloid Plaque Deposition as measured by PET Scan | baseline; 12 weeks.
Change from baseline on the Neuropaychiatic Inventory (NPI) | baseline; 6 weeks; 12 weeks; 24 weeks.
Change from baseline on the Alzheimer's Disease Cooperative study-Activities of Daily Living Scale(ADCS-ADL) | baseline; 6 weeks; 12 weeks; 24 weeks.
Change from baseline on the Alzheimer's Disease Cooperative study-clinical global impression of change scale(ADCS-CGIC) | baseline; 6 weeks; 12 weeks; 24 weeks.
Change from baseline on the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) | baseline; 6 weeks; 12 weeks; 24 weeks.
Change from baseline on the Mini Mental state Examination (MMSE) score | baseline; 6 weeks; 12 weeks; 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, Study Chair — M.D., Ph.D.
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No